CLINICAL TRIAL: NCT03610165
Title: The Role of Acumen Hypotension Prediction Index Software in Hypotension Management During Moderate to High-Risk Noncardiac Surgery: A Pilot Randomized Control Trial
Brief Title: Hypotension Prediction Index for Blood Pressure Management
Acronym: HPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kamal Maheshwari, MD MPH, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-557
Record Dates: First submitted 2018-07-13; First posted 2018-08-01 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Intraoperative Hypotension

STUDY DESIGN:
Intervention Model Description: Single-center randomized comparison of invasive arterial pressure monitoring vs. arterial pressure monitoring combined with Acumen Hypotension Prediction Index (HPI) software guidance on intraoperative hypotension duration and severity.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arterial line - Control (Placebo Comparator): Arterial line waveform and pressure
  Interventions: Device: Control
- Acumen HPI-enabled EV1000 screen (Experimental): Arterial line waveform and pressure + HPI alert from EV1000 monitor
  Interventions: Device: Acumen HPI-enabled EV1000 screen

INTERVENTIONS:
Device: Acumen HPI-enabled EV1000 screen — Acumen HPI-enabled EV1000 screen.
  Arms: Acumen HPI-enabled EV1000 screen
Device: Control — Arterial waveform and pressures
  Arms: Arterial line - Control

SUMMARY:
Design: Single-center randomized comparison of invasive arterial pressure monitoring vs. arterial pressure monitoring combined with Acumen Hypotension Prediction Index (HPI) software guidance on intraoperative hypotension duration and severity.

Aim: To determine whether use of Acumen HPI software guidance to guide intraoperative hemodynamic management in the non-cardiac surgery reduces the duration and severity of hypotension.

Primary hypothesis: Our primary hypothesis is that adding Acumen HPI software guidance to the information provided by the invasive arterial pressure monitoring during moderate- to high-risk noncardiac surgery reduces time-weighted average (TWA) intraoperative hypotension below a threshold of 65 mmHg.

DETAILED DESCRIPTION:
STUDY RATIONALE Even when clinicians try to prevent intraoperative hypotension, they often fail because it is difficult to predict which patients will become hypotensive, much less when. A risk score for predicting minute-by-minute intraoperative hypotension is not currently available. Yet it seems likely that ability to identify when a patient is likely to become hypotensive, and the pathophysiology of the event, will improve hemodynamic management and perhaps patient outcome. Acumen HPI appears to be a reliable predictor of intraoperative hypotension, and should thus help clinicians anticipate and avoid hypotension. Furthermore, the secondary guidance provided by the Acumen HPI may help clinicians optimally manage fluids and thus prevent future episodes in the same patient.

AIMS To determine whether use of Acumen HPI software to guide intraoperative hemodynamic management in the non-cardiac surgery reduces the duration and severity of hypotension.

PRIMARY HYPOTHESIS Our primary hypothesis is that use of the Acumen HPI software guidance reduces TWA intraoperative hypotension below a threshold of 65 mmHg.

Specifically, we will compare the amount of intraoperative hypotension below mean-arterial pressure (MAP) threshold of 65 mmHg, in patients randomized to invasive arterial pressure monitoring vs. invasive arterial pressure monitoring with Acumen Hypotension Prediction Index software. In both cases, clinicians will strive to keep MAP above 65 mmHg to the extent practical.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥45 years
* ASA Physical Status 3 or 4
* Moderate- or high-risk surgery (for example, orthopedic, spine, urology, and general surgery)
* Planned invasive blood pressure monitoring
* General anesthesia
* Surgery duration expected to last >2 hours
* Planned overnight hospitalization

Exclusion Criteria:

* Contraindication to the invasive blood pressure monitoring
* Pregnancy
* Emergency surgery
* Known clinically important intracardiac shunts
* Known aortic stenosis with valve area ≤ 1.5 cm2
* Known moderate to severe aortic regurgitation
* Known moderate to severe mitral regurgitation
* Known moderate to severe mitral stenosis
* Patient or surgical procedure type known as an SVV limitation16 (e.g. tidal volume <8mL/kg of theoretical ideal weight, spontaneous ventilation, persistent cardiac arrhythmia, known atrial fibrillation, open chest surgery, Heart Rate/Respiratory Rate (HR/RR) ratio <3.6)
* Current persistent atrial fibrillation
* Congestive heart failure with ejection fraction <35%
* Neurosurgery
* Emergent or cardiovascular surgical procedure
* Patient who is confirmed to be pregnant
* Refusal of patient or authorized representative to sign consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Maheshwari, MD, MPH, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Maheshwari K, Shimada T, Fang J, Ince I, Mascha EJ, Turan A, Kurz A, Sessler DI. Hypotension Prediction Index software for management of hypotension during moderate- to high-risk noncardiac surgery: protocol for a randomized trial. Trials. 2019 May 3;20(1):255. doi: 10.1186/s13063-019-3329-0. PMID 31053082

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 214 met inclusion criteria and were randomized to treatment. One patient was excluded from analysis due to non-availability of data from technical issues.
Period: Overall Study
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Started | 108 | 106
Completed | 108 | 105
Not Completed | 0 | 1
Not completed — Device didn't work | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen | Total
Number analyzed (Participants) | 108 | 105 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10) | 67 (10) | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 47 | 90
  Male | 65 | 58 | 123
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time- Weighted Average (TWA) MAP Under a Threshold of 65 mmHg.
Description: MAP stands for mean arterial pressure. Time-weighted average MAP below 65 mmHg threshold for each patient was derived by dividing AUC-MAP by the time interval between the first and the last MAP measurements.
Time Frame: MAP measurements were recorded every 20 s by the EV1000 system from induction (start anesthesia) to leaving Operation room (end of surgery).
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Number analyzed (Participants) | 108 | 105
mmHg | 0.14 [0.03 to 0.39] | 0.14 [0.03 to 0.37]
Statistical Analysis 1: Comparison: Arterial Line - Control vs Acumen HPI-enabled EV1000 Screen; Test type: Superiority; p = 0.757, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-0.03 to 0.04]

2. Primary Outcome: Hypotension Severity (AUC-MAP) Under a Threshold of 65.
Description: MAP stands for mean arterial pressure; Calculation of a specific area started when MAP was less than 65 mmHg and ended when MAP was greater than 65 mmHg; Hypotension severity (AUC-MAP) below the threshold of 65 mmHg was calculated as the cumulative sum of the areas below the given threshold for a patient using the trapezoid rule and measured in units of mmHg times minutes.
Time Frame: MAP measurements were recorded every 20 s by the EV1000 system from induction (start anesthesia) to leaving Operation room (end of surgery) .
Measure: Median (Inter-Quartile Range); unit: mmHg·min
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Number analyzed (Participants) | 108 | 105
mmHg·min | 34.2 [8.5 to 112.7] | 32.7 [6.3 to 102.0]
Statistical Analysis 1: Comparison: Arterial Line - Control vs Acumen HPI-enabled EV1000 Screen; Test type: Superiority; p = 0.715, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.3, 95% CI 2-sided [-12 to 7]

3. Primary Outcome: Duration of MAP Under a Threshold of 65 mmHg.
Description: MAP stands for mean arterial pressure; Duration is the total amount of time (in minutes) that the MAP under a threshold of 65 mmHg
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Number analyzed (Participants) | 108 | 105
min | 9.3 [2.3 to 23.5] | 7.7 [2.0 to 18.3]
Statistical Analysis 1: Comparison: Arterial Line - Control vs Acumen HPI-enabled EV1000 Screen; Test type: Superiority; p = 0.328, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1, 95% CI 2-sided [-3.3 to 1]

4. Secondary Outcome: Time-weighted Average MAP Below a Threshold of 60 mmHg Per Case
Description: MAP stands for mean arterial pressure. Time-weighted average MAP below 60 mmHg threshold for each patient was derived by dividing AUC-MAP by the time interval between the first and the last MAP measurements.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Number analyzed (Participants) | 108 | 105
mmHg | 0.02 [0.00 to 0.11] | 0.03 [0.00 to 0.13]
Statistical Analysis 1: Comparison: Arterial Line - Control vs Acumen HPI-enabled EV1000 Screen; Test type: Superiority; p = 0.376, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-0.001 to 0.011]

5. Secondary Outcome: Time-weighted Average MAP Below a Threshold of 55 mmHg Per Case
Description: MAP stands for mean arterial pressure. Time-weighted average MAP below 55 mmHg threshold for each patient was derived by dividing AUC-MAP by the time interval between the first and the last MAP measurements.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Number analyzed (Participants) | 108 | 105
mmHg | 0 [0 to 0.03] | 0 [0 to 0.04]
Statistical Analysis 1: Comparison: Arterial Line - Control vs Acumen HPI-enabled EV1000 Screen; Test type: Superiority; p = 0.226, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]

6. Secondary Outcome: Hypotension Severity (AUC-MAP) Under a Threshold of 60 mmHg.
Description: MAP stands for mean arterial pressure; Calculation of a specific area started when MAP was less than 60 mmHg and ended when MAP was greater than 60 mmHg.
  Hypotension severity (AUC-MAP) below the threshold of 60 mmHg was calculated as the cumulative sum of the areas below the given threshold for a patient using the trapezoid rule and measured in units of mmHg times minutes.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg·min
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Number analyzed (Participants) | 108 | 105
mmHg·min | 5.3 [0.00 to 29.2] | 6.0 [0.33 to 28.3]
Statistical Analysis 1: Comparison: Arterial Line - Control vs Acumen HPI-enabled EV1000 Screen; Test type: Superiority; p = 0.610, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-0.67 to 2.00]

7. Secondary Outcome: Hypotension Severity (AUC-MAP) Under a Threshold of 55 mmHg.
Description: MAP stands for mean arterial pressure; Calculation of a specific area started when MAP was less than 55 mmHg and ended when MAP was greater than 55 mmHg.
  Hypotension severity (AUC-MAP) below the threshold of 55 mmHg was calculated as the cumulative sum of the areas below the given threshold for a patient using the trapezoid rule and measured in units of mmHg times minutes.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg·min
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Number analyzed (Participants) | 108 | 105
mmHg·min | 0.17 [0 to 6.7] | 1.00 [0 to 7.7]
Statistical Analysis 1: Comparison: Arterial Line - Control vs Acumen HPI-enabled EV1000 Screen; Test type: Superiority; p = 0.302, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]

8. Secondary Outcome: Duration of MAP Under a Threshold of 60 mmHg.
Description: MAP stands for mean arterial pressure; Duration is the total amount of time (in minutes) that the MAP under a threshold of 60 mmHg
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Number analyzed (Participants) | 108 | 105
min | 2.0 [0.00 to 7.7] | 2.0 [0.33 to 7.3]
Statistical Analysis 1: Comparison: Arterial Line - Control vs Acumen HPI-enabled EV1000 Screen; Test type: Superiority; p = 0.889, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-0.67 to 0.67]

9. Secondary Outcome: Duration of MAP Under a Threshold of 55 mmHg.
Description: MAP stands for mean arterial pressure; Duration is the total amount of time (in minutes) that the MAP under a threshold of 55 mmHg.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
Number analyzed (Participants) | 108 | 105
min | 0.17 [0 to 1.7] | 0.67 [0 to 2.3]
Statistical Analysis 1: Comparison: Arterial Line - Control vs Acumen HPI-enabled EV1000 Screen; Test type: Superiority; p = 0.403, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]

ADVERSE EVENTS:
Time Frame: During the hospital stay. The median length of hospital stay of both groups is 6 days.
Arm/Group | Arterial Line - Control | Acumen HPI-enabled EV1000 Screen
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/105
Other Adverse Events (participants affected / at risk) | 0/108 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT03610165/Prot_SAP_000.pdf